CLINICAL TRIAL: NCT02211443
Title: A Phase I Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of SCT200, a Recombinant Full Human Anti-epidermal Growth Factor Receptor(EGFR) Monoclonal Antibody，in Patients With Metastatic Colorectal Cancer Following Fluoropyrimidine, Irinotecan and Oxaliplatine Chemotherapy Regiment
Brief Title: Safety, Tolerability and Pharmacokinetics of Recombinant Anti-epidermal Growth Factor Receptor(EGFR) Monoclonal Antibody in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCT200mCRCI
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Full human anti-EGFR monoclonal antibody (SCT200) ;; metastatic colorectal cancer （mCRC）;; Escalating doses ;; single dose and multiple doses;; safety, tolerability and pharmacokinetics.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Two phase study of Recombinant full human Anti-epidermal growth factor receptor(EGFR) Monoclonal Antibody:
  First phase: seven escalating single-dose groups : 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0 mg/kg
  Second phase: multiple-dose groups 0.5, 1.0, 2.0, 3.0 mg/kg: weekly once for 4 doses; 5.0, 6.0 mg/kg: every two weeks for 2 doses; 4.0 mg/kg: weekly or every two weeks depends on the results of previous dose groups.
  Interventions: Biological: Recombinant full human Anti-EGFR Monoclonal Antibody

INTERVENTIONS:
Biological: Recombinant full human Anti-EGFR Monoclonal Antibody
  Other Names: SCT200

SUMMARY:
The purpose of this study is to determine whether SCT200 is safe and tolerant in the treatment of metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 70 years;
* having histologically confirmed metastatic colorectal cancer;
* having experienced previous treatment failures including fluoropyrimidine, irinotecan and oxaliplatine chemotherapy regiment;
* having determined wild-type KRAS tumor;
* having to have measurable or nonmeasurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; and expected survival of at least ≥3 months;
* adequate hematological, renal and liver functions:

  1. Hematological function: white blood cell count of >4.0×109/L; absolute neutrophil count of >1.5×109/ L; platelet count of >100×109/L; hemoglobin level of >90.0 g/L;
  2. Renal function: serum creatinine level of<1.5×upper limit of normal (ULN);
  3. Liver function: total bilirubin level of<1.5×ULN; aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of <1.5×ULN; or <5 × ULN for patients with liver metastases;
* no other malignancies only if they had following malignancies , which were not required to treat or who had curative resection: cervical carcinoma in situ, the skin basal carcinoma or squamous cell carcinoma, bladder epithelial tumors, or only they had some malignancies requirement only surgical therapy and disease free survival≥5 years;
* no serious nonmalignant diseases including hypertension, diabetes mellitus, coronary artery disease, and mental disorder.
* not pregnant; or not lactating; or accepted birth control methods during the study;
* signed an informed consent form which was approved by the institutional review board of the respective medical center .

Exclusion Criteria:

* had received EGFR target treatment including EGFR tyrosine kinase inhibitors(TKI), or anti- EGFR monoclonal antibody;
* having to be at least 4 weeks beyond prior anticancer therapy (including corticosteroid , or nitrosourea or mitomycin within 6 weeks of study entry) or participating in other clinical trial, or have not recovered from significant toxicities of prior therapy;
* chronic use of medication that could interfere with the assessment of drug-related toxicities or immunologic activity (high dose prednisone or high dose non-steroid anti-inflammatory medication);
* had recent major surgery (within 28 days);
* with symptomatically brain metastases (with the exception of clinically brain metastases stable and of no requirement further treatment);
* with active infection requirement systemic antibiotics treatment; or serious cardiovascular disease;or with evidence of active hepatitis B or C infection; or with human immunodeficiency virus infection;
* had acute pulmonary disorder; or interstitial pneumonia; or symptomatically chronic obstructive pulmonary disease (COPD) or with risk factors to COPD;
* with eye inflammation or infection, or any risk factors who could lead to eye disease;
* with a history of allergic reaction or protein product allergy including antibodies product;
* pregnant, or lactating, or not accepted birth control methods including male patients.
* had a history of alcohol or drugs addiction, or with any risk which may affect the patient's health evaluation or mantle state

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with SCT200-related adverse events | up to 105 days

SECONDARY OUTCOMES:
Area Under the plasma concentration versus time curve (AUC) of SCT200 | prior to the initial dose and 0,0.5,1,2,4,8,24,48 hours,4,7,14,21days post- first dose

OTHER OUTCOMES:
Time to Disease Progression (TTP) of SCT200 | up to 105 days

REFERENCES:
- [Derived] Zhang W, Han X, Yang L, Song Y, Xie L, Gai W, Wang Y, Shi Y. Safety, pharmacokinetics and efficacy of SCT200, an anti-EGFR monoclonal antibody in patients with wild-type KRAS/NRAS/BRAF metastatic colorectal cancer: a phase I dose-escalation and dose-expansion study. BMC Cancer. 2022 Oct 28;22(1):1104. doi: 10.1186/s12885-022-10147-9. PMID 36307775